CLINICAL TRIAL: NCT02502643
Title: The Efficacy of OK-432 Pleurodesis on Postoperative Air Leak
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201504066RINA
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Postoperative Air Leak
Keywords: Safety and Efficacy; Thoracic Surgery
MeSH Terms: interventions — Picibanil; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OK-432 pleurodesis (Experimental): Picibanil ( OK-432 ) ,OK-432 (KE Z Klinische Einbeit; 1 KE contains 0.1 mg of dried cocci; UKIMA PLANT OF CHUGAI PHARMA MANUFACTURING CO, LTD; JAPAN).
  Interventions: Drug: OK-432 pleurodesis
- normal saline pleurodesis (Active Comparator): (Normal Saline),Isotonic Sodium Chloride Solution
  Interventions: Drug: normal saline pleurodesis

INTERVENTIONS:
Drug: OK-432 pleurodesis — 1.Pain medications (if no contraindications) Before half hour; Bain (IM ,0.15mg / kg). 2. Make the patient supine position 3. Near the body of patient's chest tube is the injection site disinfection with the alcoholic Betadine and alcohol repeated three times.4. 20 cc of 2% lidocaine hydrochloride (400 mg) was instilled into the pleural cavity through the chest tube 5. A solution of 30 cc of normal saline containing 5 KE of OK-432 (KE Z Klinische Einbeit; 1 KE contains 0.1 mg of dried cocci).6. Inject air 20 cc 7. The injection site will cover with op site and the rubber tube that connecting the chest tube and chest bottle was raised 40-60 cm above the patient to trap the sclerosing agent but allow air to pass 8. Patients will reposition (left and right side)every 30 minutes in 2 hours
  Other Names: Picibanil
  Arms: OK-432 pleurodesis
Drug: normal saline pleurodesis — Make the patient supine position , Near the body of patient's chest tube is the injection site disinfection with the alcoholic Betadine and alcohol repeated three times.injected a solution of 30 cc of normal saline , and then injected into 20 cc air to the rubber chest tube , so that normal saline can completely into the chest, the injection site will cover with op site, use a rubber band to the rubber chest tube for hanging from the patient's body 40-60 cm high.Patients will reposition (left and right side)every 30 minutes in 2 hours
  Other Names: normal saline
  Arms: normal saline pleurodesis

SUMMARY:
The purpose of this study is (1) The success rate of OK-432 pleurodesis after thoracic surgery that air leak over 48 hours (2)The side effects and treatments of OK-432 pleurodesis.

[Methods] This study was a prospective, randomized, open-label, controlled study to evaluate the effectiveness of OK-432 pleurodesis of persistent air Leak after pulmonary Resection. The adult patient have persistent air leak >48 hours after thoracic surgery, will randomized to OK-432 pleurodesis (OK-432 group) or normal saline pleurodesis (NS group). The trial will be conduct from May 25, 2015 to May 25, 2018 in the Department of Surgery at national Taiwan University Hospital, a medical center. The study protocol was approved by the hospitals' Institutional Review Boards. A total of 80 cases, the subjects will be the hospital thoracic surgery ward and received outpatient programs. Eligible Subjects : adults (minimum age> 20 years; maximum age ≦ 70 years old) patients with thoracic surgery and over48 hours of continuous air leak. The exclusion criteria include: penicillin allergy,primary pneumothorax, esophageal cancer, immune dysfunction, those who can not sign a consent form, and pregnant or lactating, other serious concomitant illness such as uremia or liver cirrhosis. Study steps: eligible Patients will randomize according to computer-generated random numbers, with 1:1 ratio in sequentially numbered, sealed envelopes by a study nurse who was masked to the study. Randomization envelopes were opened, and randomization was performed by the study nurse after informed consent was obtain. Eligible inpatients were randomized to the OK-432 group or the normal saline (NS) group，each group are 40 cases.

All subjects were observed by the physician who was masked to the study， about air leak stop time, chest tube removal time, discharge time, outpatient chest X-ray, pulmonary function tests as necessary. cases if persistent air leak more than seven days, the attending physician determines whether pleurodesis again or surgery or other medical treatment. Finally, the researcher who do not know groups will collection data by "air leak case record form" including diagnosis, surgical site，the start and end time of the surgery, the use of antibiotics, discomfort problems (pain , stomach discomfort, cough, fever> 38 ℃, allergic reactions and respiratory discomfort), postoperative air leak time, air leak stop time , chest tube removal time, discharge time, the data will be use SPSS20.0 version of the statistical software package, and T-test, pair T-test ，Anova ,linear correlation statistical methods for analysis.

Outcome measures: OK-432 success rate, OK-432 side effects, air leak time, chest tube remove time, length of hospital stay.

DETAILED DESCRIPTION:
[Background and Objective] :Air leak produced after thoracic surgery is a common phenomenon.Prolonged chest tube placement can lead to empyema or infection, and extended hospitalization or even death. In 2010 many researchers reported that The incidence of lung resection produce air leak about 8-26% (Singhal et al., 2010), and even up to 50% (Mueller & Marzluf, 2014).How to effectively treatment is still not clear.The chemical pleurodesis is an effective option in management of air leak.There are several chemical agents for pleurodesis, such as tetracycline and minocycline, talc, Taurolidine, bleomycin, iodopovidone, picibanil (OK-432), silver nitrate, quinacrine. What kind of chemical agent effective remain controversial. A study evaluated after thoracoscopic operation for primary spontaneous pneumothorax the safety and efficacy of chemical pleurodesis with a comparison between minocycline and OK-432. The OK-432 pleurodesis (19 patients) as the primary treatment and the primary success rate was 95%.(How et al., 2014).Another retrospective case-control study examining post-isolated lobectomies and bilobectomies by thoracotomy of Persistent air leak，sclerosis (talc, bleomycin, minocycline, doxycycline)for the treatment of prolonged air leak was successful in 40 of 41 patients (the success rate of 97.6%) (Liberman et al., 2010). The prolonged air leaks after major pulmonary resection still no empirical treatment of clinical research.

Hypothesis: patients were persistent air leak after 48 hours chest surgery will perform OK-432 pleurodesis .The chest tube time can reduce and length of hospital stay. Extended applications can significantly reduce medical costs and manpower, and to explore OK -432 pleurodesis side effects and treatment.

ELIGIBILITY:
Inclusion criteria:

* Patients were eligible for this study if they were more than 20 and less than 70 years old of age and under thoracic surgery that air leak lasting more than 48 hours form chest drainage bottles.

Exclusion criteria :

* penicillin allergy, primary pneumothorax, esophageal cancer, immune dysfunction, those who can not sign a consent form, and pregnant or lactating, other serious concomitant illness such as uremia or liver cirrhosis.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
OK-432 success rate | 48 hours
  The success rate of OK-432 was defined chest bottle no bubbles appear when coughing, then CXR was perform the next day after pleurodesis, and after cessation of the air leak,the chest tube is remove .

SECONDARY OUTCOMES:
OK-432 side effects | 48 hours
  The main side effects of the procedure with OK-432 were fever and chest pain, which were well controlled by non-steroidal anti-inflammatory drugs.the side effects of OK-432 will be assessed by temperature,visual analog scale.these will present as number and frequencies (%).

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Test2, Taiwan